CLINICAL TRIAL: NCT03688373
Title: Optimizing Exposure in the Treatment of Anxiety in Youth: Facing Fears in Big or Smalls Steps?
Brief Title: Facing Fears in Big or Smalls Steps?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Rachel de Jong, PhD Student, University of Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL59986.042.16
Record Dates: First submitted 2018-07-30; First posted 2018-09-28 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Specific Phobia
MeSH Terms: conditions — Phobia, Specific | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure-in-big-steps (Experimental): In the big steps exposure sessions the adolescent moves in three a set pace of big steps from bottom to top (1-5-10) in their fear hierarchy. From 0-5 in the first session and from 5-10 in the second session.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Exposure-in-small-steps (Experimental): In the small steps exposure sessions the adolescent moves in a step-by-step pace of their own choice from bottom to top in their fear hierarchy, for example from 1 to 2 to 3 to in the first session and from 4 to 5 to 6 etc. in the second session.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Each intervention will contain a 60-minute psycho-education session (PE) and two 60-minute exposure sessions (EX), conducted by a mental health professional together with a master student in psychology, who are both weekly supervised by a CBT certified psychologist. In the first (PE) session, participants learn about anxiety, specific phobias and exposure. During this session they will create a fear hierarchy (1 relating to least fearful and 10 indicating most fearful situation), formulate their cognition about the feared object or situation and determine what they want to achieve during treatment (e.g. goal situation). The next two sessions consist of exposure exercises in either big or small steps.

SUMMARY:
Anxiety problems are a major concern of youth mental health given that the prevalence of anxiety disorders in Dutch adolescents aged 12 to 18 is approximately 10 percent. In this group, specific phobias are among the most common. Cognitive Behavioral Therapy (CBT) with exposure as its key ingredient, takes a prominent place in national guidelines for the treatment of anxiety disorders. These guidelines are based on empirical support that exposure is effective in the treatment of specific phobia. Therapists help phobic adolescents to overcome their fear by gradually, step by step, working their way up from less scary situations to situations that cause a greater deal of anxiety. Although it is clear that exposure is effective, the size of the steps to be taken in this process remains unclear. However, there are multiple reasons to assume that one or the other works best. On the one hand, adolescents will soon gain trust in their own abilities when taking small steps, which enlarges their feeling of self-control (e.g., self-efficacy). On the other hand there is the risk that these small steps might be experienced as safety behavior and avoidance, which is counterproductive to the essence of exposure (i.e., overcoming the fear) and undermines the potential effect. This might result in either a longer treatment or insufficient treatment benefits. Considering this risk, and the fact that confrontation with a feared object or situation in daily life is also not a step-by-step process, this study proposes to evaluate the optimal dosage of exposure, by studying whether exposure in big steps is more effective than exposure in small steps.

DETAILED DESCRIPTION:
Objective: The primary goal of this study is to evaluate whether exposure in big steps is more effective than a small step-by-step approach. The secondary goal is to find child, parent and therapist factors that possibly relate to the effectiveness of the exposure exercises.

Study design: Randomized Controlled Trial (RCT) with two parallel groups (intervention versus intervention).

Study population: Adolescents aged 12 to 17 years with a specific phobia of the animal/situational subtype.

Intervention (if applicable): The intervention will be designed as a CBT, a therapy which has proven to be effective in treating specific phobia. The intervention consists of three individual sessions, each up to 60 minutes long. Each condition starts with a psycho-education session on specific phobias and exposure, during which the participants will create a fear hierarchy (from 1 as least fearful to 10 as most fearful). Following this session either two exposure-in-big-steps or two exposure-in-small-steps sessions are offered. In the big steps exposure condition the adolescent moves in three big steps from bottom to top (1-5-10) in their fear hierarchy. In the small steps exposure condition the adolescent moves in many small steps from bottom to top in their fear hierarchy, for example from 1 to 2 to 3 to 4 etc. The intervention will be provided by an experienced mental health professional.

Main study parameters/endpoints (see outcome measures paragraph): The main study parameter isseverity of the specific phobia. Secondary study parameters are out-session fear, fearful cognitions, bodily tension, avoidance, coping, in-session fear, in-session harm expectancy (possible mediator variables), approach behavior and self-efficacy. Tertiary study parameters are healthcare costs and quality of life (cost-effectiveness), note: cost-effectiveness is assessed for another study. Other study parameters are specific phobiadiagnosis, general comorbidity, comorbid anxiety and depression, and demographic variables (possible moderator variables); and credibility and expectancy of the treatment, treatment satisfaction, treatment integrity and therapeutic alliance (treatment characteristics).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12-17 years old and in secondary school
* Sufficient knowledge of the Dutch language
* Meeting the criteria of specific phobia of the situational or animal subtype

Exclusion Criteria:

* Absence of permission of legal guardian(s)
* Currently in treatment or receiving medication for anxiety
* Received CBT for anxiety in the past 12 months
* Specific phobia that do not fall under the situational or animal subtype, for example:

  * Aerophobia: fear of flying
  * Emetophobia: fear of vomiting
  * Hemophobia: fear of blood
  * Hosophobia: fear of infection
  * Astraphobia: fear of lightning
* Different and more urgent request for help
* (Risk of) suicidality, psychosis or domestic violence

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Change in specific phobia severity (Interference, number of symptoms and general impression of the psychologist) | Time Frame: At intake (T0), four weeks later at pre-intervention assessment (T1), another four weeks later at post-intervention assessment (T5) and another four weeks later at follow-up assessment (T6)
  Specific phobia severity in children will be measured with a clinical semi-structured interview using the Anxiety Disorder Interview Schedule for Children and Parents (ADIS-IV-C/P). The study will only include the section of specific phobia. Severity of the specific phobia will be rated on a 0-8 interval scale by an independent psychologist on the ADIS-IV (see above). This rating is based on the level of interference, number of symptoms and general impression of the psychologist. A rating 0, 1, 2 or 3 is labelled as no specific phobia, a rating of 4 or 5 is labelled as a mild specific phobia, whereas a rating of 6, 7 or 8 means the specific phobia is labelled as severe. This rating is used to randomize the participants to the different conditions. The ADIS-IV has good test-retest reliability and concurrent validity.

SECONDARY OUTCOMES:
Change in level of anxiety (Subjective level of fear, Fearful cognitions, Bodily tension, Avoidance and Coping) | Time Frame: In the first treatment session (T2), one week later in the second treatment session (T3), one week later in the third treatment session (T4), and one week later at post-intervention (T5), and four weeks later at follow-up assessment (T6)
  Level of anxiety compromised of Subjective level of fear, Fearful cognitions, Bodily tension, Avoidance and Coping will be measured by Visual Analogue Scales (VAS) ranging from 0-100 (ratio scale) on which the child rates the following aspects of the goal situation as set in the PE session:
  * Subjective level of fear: 'Not frightened at all' (0) - 'Completely frightened' (100)
  * Fearful cognitions: 'I do not believe this at all' (0) - 'I completely believe this' (100), in which the credibility of the cognition about the feared object or situation as set in the PE session is rated.
  * Bodily tension: 'My body feels not tense at all' (0) - 'My body feels completely tense' (100)
  * Avoidance: 'I would never avoid this situation/object if I could' (0) - 'I would always avoid this situation/object if I could' (100)
  * Coping: 'I cannot cope with this situation/object at all when I encounter it' (0) - 'I can completely cope with this situation/object when I encounter it' (100)
Change in approach behaviour (Time and Distance) | Time Frame: At pre-intervention assessment (T1), four weeks later at post-intervention assessment (T5) and four weeks later at follow-up assessment (T6)
  Approach behaviour will be measured by three situational Behavioural Approach Tests (BAT) for feared and avoided objects or situations. The test consists of a number of increasingly difficult steps in which children are asked to approach a phobic object or situation, but are told they can stop the test at any time they wish to do so. During the BAT, individuals are asked to provide "subjective unit of disturbance scale" (SUDS 0-100 ratio scale) ratings immediately after encountering the phobic animal or situation.
Change in self-efficacy (Academic, Social and Emotional) | Time Frame: At pre-intervention assessment (T1), four weeks later at post-intervention assessment (T5) and four weeks later at follow-up assessment (T6)
  Self-efficacy will be measured by the Self Efficacy Questionnaire for Children (SEQ-C). This questionnaire contains 24 questions regarding academic, social and emotional self-efficacy. Items are rated on a 5-point interval scale from 'not at all' (1) to 'very well' (5). The SEQ-C is proven to be a valid instrument with sufficient reliability.

OTHER OUTCOMES:
Cost-effectiveness (Healthcare costs and In quality adjusted life years) | Time Frame: At pre-intervention assessment (T1) and eight weeks later at follow-up assessment (T6)
  In addition, cost-effectiveness of the intervention will be assessed by measuring costs and quality of life (effectiveness). Measuring cost-effectiveness is not the primary goal of this research but since this study is part of a larger national project in which cost-effectiveness will also be taken into account, we consider it relevant to state here.
  * Healthcare costs will be measured by registration of costs in a cost diary based on the Trimbos Institute and Institute of Medical Technology Assessment Questionnaire on Costs Associated with Psychiatric Illness (TiC-P) and PRODISQ.
  * The EuroQol Questionaire (EQ-5D-Y youth version) will be used to establish quality of life as expressed in quality adjusted life years (QALYs).
  Healthcare costs and in quality adjusted life years are combined to report cost-effectiveness.
Change in specific phobia diagnosis (Interference, number of symptoms and general impression of the psychologist) | Time Frame: At intake (T0), four weeks later at pre-intervention assessment (T1), another four weeks later at post-intervention assessment (T5) and another four weeks later at follow-up assessment (T6)
  Specific phobia diagnosis will be assessed with the ADIS IV (see above). All items offer three possible answers: 'yes', 'no' or 'other' on a nominal scale (which is chosen when the adolescent answers 'I don't know' or 'sometimes'). If the adolescent meets all four criteria for specific phobia as set in the ADIS-IV, he or she can participate in the study.
Comorbid anxiety and depression symptoms | Time Frame: At pre-intervention assessment (T1), four weeks later at post-intervention assessment (T5) and another four weeks later at follow-up assessment (T6)
  Given the high comorbidity of anxiety and depression in children, comorbid anxiety and depression will be assessed with the Revised Child Anxiety and Depression Scale for Children and Parents (RCADSC/ P) consisting of 47 items and the Phobia section of the Spence Children's Anxiety Scale for Children and Parents (SCAS-C/P) consisting of 9 items. All items are rated on a 4-point interval scale from 'never' to 'always'. Both the RCADS (Chorpita, Moffitt, & Gray, 2005) and the SCAS (Whiteside & Brown, 2008) have good psychometric properties, and are combined into the RCADSCAS for this study.
Change in in-session fear before and after each exposure exercise | During the second (T3) and the third (T4) treatment session
  In-session fear is measured before and after every in-session exposure step, by asking the adolescent to provide "subjective unit of disturbance scale" (SUDS) ratings on a ratio scale 0-100 immediately before and after a new step in encountering the phobic object or situation.
In-session harm expectancy before and after each exposure exercise | During the second (T3) and the third (T4) treatment session
  In-session harm expectancy is measured before and after every in-session exposure step. Before every exposure step the adolescent is asked: a) 'What are you most worried will happen?', b) 'On a (ratio) scale 0-100, how likely does this seem?, and c) 'On a (ratio) scale 0-100, how bad would it be if the thing you are most worried about will occur?'. After every exposure step the adolescent is reminded of their worry and asked: a) 'On a (ratio) scale 0-100, how likely does it seem this would happen if we would repeat this step?', and b) 'On a (ratio) scale 0-100, how bad would it be if the thing you are most worried about will occur?'.
Change in treatment credibility and expectancy of the treatment | At pre-intervention assessment (T1), four weeks later at post-intervention assessment (T5) and another four weeks later at follow-up assessment (T6)
  Credibility and expectancy of the treatment are measured by the Credibility and Expectancy Questionnaire (CEQ-C/P). This questionnaire contains 6 items all rated on a 9-point interval scale. The psychometric properties of the scale have been qualified as good.
Change in treatment satisfaction during and after treatment | At pre-intervention assessment (T1), four weeks later at post-intervention assessment (T5) and another four weeks later at follow-up assessment (T6)
  Treatment satisfaction will be measured with the Service Satisfaction Scale (SSS). Four items are rated on a 4-point interval scale ranging from 'no, definitely not' to 'yes, definitely'. The psychometric properties of the scale have been qualified as good.
Therapeutic alliance during the treatment | One week after the last intervention week, at post-intervention assessment (T5)
  Therapeutic alliance is measured by the Therapeutic Alliance Scale for Children and Parents (TAS-C/P). Both parts consist of 12 items rated on a 4-point interval scale. The psychometric properties of the scale have been qualified as good.

CONTACTS AND LOCATIONS:
Overall Officials: Peter de Jong, Prof, Study Chair — University of Groningen; Maaike Nauta, Prof, Study Director — University of Groningen; Miriam Lommen, Dr, Study Director — University of Groningen
Locations (3):
- Netherlands (3):
  - Accare Drachten, Drachten, Provincie Friesland
  - Accare Leeuwarden, Leeuwarden, Provincie Friesland
  - Accare Universitair Centrum voor Kinder en Jeugdpsychiatrie, Groningen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Silverman WK, Saavedra LM, Pina AA. Test-retest reliability of anxiety symptoms and diagnoses with the Anxiety Disorders Interview Schedule for DSM-IV: child and parent versions. J Am Acad Child Adolesc Psychiatry. 2001 Aug;40(8):937-44. doi: 10.1097/00004583-200108000-00016. PMID 11501694
- [Background] Wood JJ, Piacentini JC, Bergman RL, McCracken J, Barrios V. Concurrent validity of the anxiety disorders section of the Anxiety Disorders Interview Schedule for DSM-IV: child and parent versions. J Clin Child Adolesc Psychol. 2002 Sep;31(3):335-42. doi: 10.1207/S15374424JCCP3103_05. PMID 12149971
- [Background] Koopmanschap MA. PRODISQ: a modular questionnaire on productivity and disease for economic evaluation studies. Expert Rev Pharmacoecon Outcomes Res. 2005 Feb;5(1):23-8. doi: 10.1586/14737167.5.1.23. PMID 19807557
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Brady EU, Kendall PC. Comorbidity of anxiety and depression in children and adolescents. Psychol Bull. 1992 Mar;111(2):244-55. doi: 10.1037/0033-2909.111.2.244. PMID 1557475
- [Background] Chorpita BF, Moffitt CE, Gray J. Psychometric properties of the Revised Child Anxiety and Depression Scale in a clinical sample. Behav Res Ther. 2005 Mar;43(3):309-22. doi: 10.1016/j.brat.2004.02.004. PMID 15680928
- [Background] Wolitzky-Taylor KB, Horowitz JD, Powers MB, Telch MJ. Psychological approaches in the treatment of specific phobias: a meta-analysis. Clin Psychol Rev. 2008 Jul;28(6):1021-37. doi: 10.1016/j.cpr.2008.02.007. Epub 2008 Mar 7. PMID 18410984
- [Background] Marks IM, Mathews AM. Brief standard self-rating for phobic patients. Behav Res Ther. 1979;17(3):263-7. doi: 10.1016/0005-7967(79)90041-x. No abstract available. PMID 526242
- [Background] Hedtke KA, Kendall PC, Tiwari S. Safety-seeking and coping behavior during exposure tasks with anxious youth. J Clin Child Adolesc Psychol. 2009 Jan;38(1):1-15. doi: 10.1080/15374410802581055. PMID 19130353
- [Background] Craske MG, Treanor M, Conway CC, Zbozinek T, Vervliet B. Maximizing exposure therapy: an inhibitory learning approach. Behav Res Ther. 2014 Jul;58:10-23. doi: 10.1016/j.brat.2014.04.006. Epub 2014 May 9. PMID 24864005